CLINICAL TRIAL: NCT06843863
Title: The Effects of Smartphone Addiction on Pinch Strength, Muscle Stiffness, and Hand and Wrist Function in Young Adults: A Cross-Sectional Study
Brief Title: The Effects of Smartphone Addiction on Pinch Strength, Muscle Stiffness, and Hand/Wrist Function in Young Adults
Status: Recruiting | Type: Observational
Sponsor: Istanbul Gelisim University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Istanbul Kent University (Other)
Responsible Party: Principal Investigator, Aysem Ecem Ozdemir, Research Assistant, Istanbul Gelisim University
Other Study IDs: IUC002
Record Dates: First submitted 2025-02-18; First posted 2025-02-25 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Smartphone Addiction
Keywords: Smartphone; Behavior; Addictive; Muscle stiffness; Musculoskeletal Pain
MeSH Terms: conditions — Internet Addiction Disorder; Behavior; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smartphone Addiction Group: Individuals classified as having smartphone addiction based on the Smartphone Addiction Scale-Short Version (SAS-SV). Participants in this group scored 31 or higher for males and 33 or higher for females on the SAS-SV, indicating problematic smartphone use that meets the threshold for addiction.
  Interventions: Other: No intervention.
- Non-Smartphone Addiction Group: Individuals who are not classified as having smartphone addiction based on the Smartphone Addiction Scale-Short Version (SAS-SV). Participants in this group scored below 31 for males and below 33 for females on the SAS-SV, indicating that their smartphone use does not meet the threshold for addiction.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — Participants allocated to the groups were assessed only once. No intervention was applied, and they were not followed up.

SUMMARY:
Smartphones have become an indispensable part of daily life, and their increasing use has raised concerns about various health effects, including musculoskeletal symptoms. Repetitive movements of the thumb and hand muscles can lead to issues such as tendinosis, myofascial pain syndrome, and a decrease in pinch strength. Studies have shown that musculoskeletal symptoms related to smartphone use are common among young adults and university students. Additionally, an increase in device size may place greater strain on the wrist and finger muscles. Repetitive movements can cause stiffness changes in the thumb muscles, and the relationship between these changes and pinch strength is considered an important research topic. In this study, we aimed to investigate the effects of smartphone addiction on pinch strength, muscle stiffness, hand/wrist pain, and function in young adults.

DETAILED DESCRIPTION:
This study was designed as a cross-sectional study. Volunteers eligible to participate were first screened based on the results of the Smartphone Addiction Scale-Short Version (SAS-SV), and they were divided into two groups as Smartphone Addiction and Non-Smartphone Addiction, with a cutoff score of 31 for males and 33 for females. Subsequently, the determination of dominant hand was performed. All assessments were conducted on the participants' dominant extremity. The assessments were carried out in the following order: Patient-Rated Wrist/Hand Evaluation Questionnaire (PRWHE), the Finkelstein test, muscle stiffness measurement, and finally, pinch strength assessment, as it was considered to potentially cause fatigue. All assessments were conducted by expert physiotherapists within a total duration of 30 minutes, and participants were not followed up afterward, nor recieved any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study
* Have been using a smartphone for more than one year
* Aged between 18 and 25 years
* Send 25 or more text messages or emails per day
* Spend more than 2 hours browsing the internet and/or play games for more than one hour a day

Exclusion Criteria:

* Having radiating/radicular pain in the upper extremity
* Having neck pain
* Congenital deformities in the upper extremity and neck
* A history of diagnosed neurological, rheumatic, musculoskeletal, or cardiovascular diseases
* Having previously undergone surgery on the neck and/or upper extremity
* Having been diagnosed with De Quervain's disease or tendinopathy in the hand/hand wrist muscles before

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University student from Istanbul Kent University and Istanbul Gelisim University.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Stiffness | Baseline
  Muscle stiffness (Abductor Pollicis Brevis, Abductor Pollicis Longus and Extensor Pollicis Brevis) was measured using the MyotonPRO (Myoton SA, Tallinn, Estonia) device. A brief mechanical impulse was applied to the muscle and then quickly released. Stiffness (N/m) is a parameter related to the capacity to withstand an external force. The reliability of the device has been proven in healthy individuals. The measurement site was marked on the skin with a pen. In all applications, the MyotonPRO probe was placed perpendicular to the skin, and in multi-scan mode, three measurements were recorded with 10 pulses at 1-second intervals. The average of the three measurements was used for analysis.
Pinch Strength | Baseline
  Lateral and palmar pinch strength were measured in kilograms using a Jamar hydraulic pinch gauge (ICC: 0.94-0.99). The measurements were performed in the standard position recommended by the American Society of Hand Therapists: seated, with the shoulder in adduction and neutral, elbow in 90 degrees of flexion, forearm in mid-rotation and supported, and wrist in neutral. Three consecutive measurements, each lasting five seconds, were taken, with one-minute rest intervals between each measurement to prevent muscle fatigue. The average of the three trials was used for analysis.

SECONDARY OUTCOMES:
Smartphone Addiction Scale-Short Version (SAS-SV) | Baseline
  The SAS-SV is a 10-item scale developed by Kwon and colleagues to measure the risk of smartphone addiction in adolescents. It is evaluated using a six-point Likert scale. The scale items are scored from 1 to 6. The scale scores range from 10 to 60, with higher scores indicating an increased risk of addiction. The scale is unidimensional and does not have subscales. In the Korean sample, the cutoff score is 31 for males and 33 for females.
Patient-Rated Wrist/Hand Evaluation Questionnaire (PRWHE) | Baseline
  This form consists of two subscales: a pain subscale with five items, a specific function subscale with six items, and a daily function subscale with four items. Each item is scored on a scale from 0 to 10. In this scale, pain and function problems are weighted equally, and the total score is measured out of 100 points.
Finkelstein Test | Baseline
  The Finkelstein test, one of the most commonly preferred clinical examination tests for diagnosing De Quervain's disease, was used. Participants were asked to make a fist with their thumb inside, and the researcher passively deviated the fist ulnarly. The presence of tenderness and pain at the radial styloid indicated a positive test.
Smartphone Surface Area | Baseline
  The dimensions of the smartphones used by the participants were measured by the researchers. Using a measuring tape, the width and length of the smartphone were recorded in centimeters. The value used for statistical analysis was determined as the surface area of the smartphone (width × length).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Kent University, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No